CLINICAL TRIAL: NCT06886854
Title: Evaluation of the Impact of Rotating Posterior and Transverse Presentations At 2 Hours of Full Dilation
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5373
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Fetus in Posterior or Transverse Position; Manual Rotation ; Obstetrics ; Delivery Room Practice
MeSH Terms: interventions — Delivery, Obstetric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Success of the rotation: Patients in labor with a fetus in posterior or transverse position at 2 hours of full dilation, verified by ultrasound. Manual rotation by an obstetrician after confirming effective analgesia, an empty bladder, and normal fetal heart rate. Success of the manual rotation
  Interventions: Device: Mode of delivery

INTERVENTIONS:
Device: Mode of delivery — Retrieval of delivery data, typically recorded by midwives - retrieval of data per delivery and post-delivery - Consultation of medical data on labor duration, labor onset method, estimated fetal weight, etc.
  Data collected for each delivery, identical in both groups.

SUMMARY:
During labor, 20% of fetuses present in a posterior or transverse position. Among them, 90% rotate spontaneously during labor. For the remaining 10%, maintaining a posterior or transverse position leads to longer labor, increased instrumental deliveries, more cesarean sections, and more severe perineal tears. Obstetricians can intervene by manually rotating the fetus to an anterior position. Several studies have shown the benefits of this technique, but they were all conducted at full dilation or one hour after full dilation. This timing does not allow enough time for the fetus to rotate spontaneously. Additionally, manual rotation can be poorly tolerated by the patient, especially if pain management is insufficient.

Our study aims to demonstrate the benefits of manual rotation two hours after full dilation. This delay allows 90% of fetuses to rotate spontaneously, and it could help harmonize obstetrical practices.

ELIGIBILITY:
Inclusion Criteria:

* - Patient delivering at Hospices Civils de Lyon (XR, HFME, LS?)
* Low-pitched voice agreement
* Mobile fetal cephalic presentation
* Transverse or posterior presentation confirmed by ultrasound
* 2 hours of complete dilation
* Agreement for 3 hours by OB-GYN
* Normal fetal heart rate
* Epidural anesthesia in place
* Bladder catheterized

Exclusion Criteria:

* - Multiparous uterus with scars
* Breech presentation
* Fetus > 5000 g
* Patient refusal
* Inadequate analgesia
* Fetal hypoxia

Ages: 15 Years to 50 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Woman in labor, not delivered at 2 hours of complete dilation, with a posterior or transverse fetal presentation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of eutocic deliveries | Collected at the time of delivery.
  Collection of delivery data recorded by the midwife: eutocic delivery, instrumental extraction by vacuum, instrumental extraction by forceps, instrumental extraction by spatula, emergency cesarean section (green, orange, or red code).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital de la croix rousse, France
  - Hopital Femme Mere Enfant, France